CLINICAL TRIAL: NCT02344472
Title: DETECT V / CHEVENDO A Multicenter, Randomized Phase III Study to Compare Chemo- Versus Endocrine Therapy in Combination With Dual HER2-targeted Therapy of Herceptin® (Trastuzumab) and Perjeta® (Pertuzumab) Plus Kisqali® (Ribociclib) in Patients With HER2 Positive and Hormone-receptor Positive Metastatic Breast Cancer.
Brief Title: Detect V / CHEVENDO (Chemo vs. Endo)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Collaborators: Roche Pharma AG (Industry); Novartis Pharmaceuticals (Industry); Eisai GmbH (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, Director Department of Obstetrics and Gynecology, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-V; 2014-002249-22 (EudraCT Number)
Record Dates: First submitted 2015-01-11; First posted 2015-01-26 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC; HER2; CTC; endocrine therapy; Pertuzumab; Trastuzumab; HER2 therapy; Ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Capecitabine; Paclitaxel; Vinorelbine; Docetaxel; exemestane; Letrozole; Anastrozole; Fulvestrant; ribociclib; 130-nm albumin-bound paclitaxel; eribulin; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Chemotherapy with docetaxel (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus docetaxel. Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Docetaxel
- Chemotherapy with paclitaxel (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus paclitaxel.Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Paclitaxel
- Chemotherapy with vinorelbine (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus vinorelbine. Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Vinorelbine
- Chemotherapy with capecitabine (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus capecitabine. Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Capecitabine
- endocrine therapy with exemestane (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus exemestane.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Exemestane; Drug: Ribociclib
- endocrine therapy with fulvestrant (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus fulvestrant.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Fulvestrant; Drug: Ribociclib
- endocrine therapy with anastrozole (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus anastrozole.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Anastrozole; Drug: Ribociclib
- endocrine therapy with letrozole (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus letrozole.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Letrozole; Drug: Ribociclib
- Chemotherapy with nab-Paclitaxel (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus nab-Paclitaxel. Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: nab-Paclitaxel
- Chemotherapy with eribulin (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus eribulin. Up to three weeks after completion of chemotherapy, patients will be treated with maintenance endocrine therapy plus dual HER2-targeted therapy and Kisqali® (Ribociclib).
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: eribulin
- endocrine therapy with leuprorelin (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus leuprorelin.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Ribociclib; Drug: leuprorelin
- endocrine therapy with goserelin (Experimental): dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (Ribociclib) plus goserelin.
  Interventions: Drug: pertuzumab; Drug: Trastuzumab; Drug: Ribociclib; Drug: goserelin

INTERVENTIONS:
Drug: pertuzumab — HER2 targeted Therapy
  Other Names: Perjeta®
Drug: Trastuzumab — HER2 targeted Therapy
  Other Names: Herceptin®
Drug: Capecitabine — Chemotherapy
  Arms: Chemotherapy with capecitabine
Drug: Paclitaxel — Chemotherapy
  Arms: Chemotherapy with paclitaxel
Drug: Vinorelbine — Chemotherapy
  Arms: Chemotherapy with vinorelbine
Drug: Docetaxel — Chemotherapy
  Arms: Chemotherapy with docetaxel
Drug: Exemestane — endocrine therapy
  Arms: endocrine therapy with exemestane
Drug: Letrozole — endocrine therapy
  Arms: endocrine therapy with letrozole
Drug: Anastrozole — endocrine therapy
  Arms: endocrine therapy with anastrozole
Drug: Fulvestrant — endocrine therapy
  Arms: endocrine therapy with fulvestrant
Drug: Ribociclib — CDK 4/6 inhibitor
  Other Names: Kisqali®
  Arms: endocrine therapy with anastrozole; endocrine therapy with exemestane; endocrine therapy with fulvestrant; endocrine therapy with goserelin; endocrine therapy with letrozole; endocrine therapy with leuprorelin
Drug: nab-Paclitaxel — chemotherapy
  Arms: Chemotherapy with nab-Paclitaxel
Drug: eribulin — chemotherapy
  Arms: Chemotherapy with eribulin
Drug: leuprorelin — endocrine therapy
  Arms: endocrine therapy with leuprorelin
Drug: goserelin — endocrine therapy
  Arms: endocrine therapy with goserelin

SUMMARY:
Chemo- versus endocrine therapy in combination with dual HER2-targeted therapy of Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus Kisqali® (ribociclib) in patients with HER2 positive and hormone-receptor positive metastatic breast cancer.

DETAILED DESCRIPTION:
Especially for diseases that are not curable such as metastatic breast cancer (MBC), the maintenance of quality of life is one of the main aims of treatments. Adverse events are well-known side effects of any cytostatic treatment and impact the patients' quality of life. Therefore, new treatment options are developed that should stop or at least slow down metastatic spread of cancer without causing negative side effects in terms of high-grade adverse events. For patients with hormone-receptor positive and HER2 positive MBC the combination of HER2-targeted therapy with endocrine therapy has already been proven to be an effective and in many cases valuable alternative to the combination of HER2-targeted therapy with chemotherapy. The high relevance of HER2-neu-targeted/endocrine treatment combinations derives from the fact that potential chemotherapy-related toxicity can be avoided, which in turn positively affects quality of life. Clinical trials suggest an additional benefit when a CDK4/6 inhibitor is added to the combination of endocrine therapy and anti HER2 treatment. DETECT V is a randomized phase III study comparing the safety and efficacy of trastuzumab plus pertuzumab and the CDK 4/6 inhibitor ribociclib in combination with either endocrine therapy or chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Signed, written informed consent in study participation
* The primary tumor and/or biopsies from metastatic sites or locoregional recurrences have been confirmed as HER2-positive (FISH-positive or IHC 3+) and hormone receptor positive breast cancer by histopathology according to local testing
* Metastatic breast cancer or locally advanced BC, which cannot be treated by surgery or radiotherapy only
* Pre- and postmenopausal women are allowed
* No more than two prior chemotherapies for metastatic disease
* No more than two prior anti-HER2 therapies for metastatic disease
* Pertuzumab retreatment is allowed if prior pertuzumab treatment was finished 12 months before
* At least one measurable lesion assessable using standard techniques by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
* Tumor evaluation according to RECIST version 1.1 has been performed within 4 weeks before randomization based on local assessment
* Age ≥ 18 years
* Standard 12-lead ECG values assessed by the local laboratory:

  * QTcF interval at screening < 450 msec (using Fridericia's correction)
  * Resting heart rate 50-90 bpm
* Left ventricular cardiac ejection fraction (LVEF) ≥ 50% at baseline (as measured by echocardiogram)
* ECOG Score ≤ 2
* Adequate organ function within 14 days before randomization, evidenced by the following laboratory results below:

  * absolute neutrophil count ≥ 1500 cells/µL,
  * platelet count ≥ 100000 cells/µL,
  * hemoglobin ≥ 9 g/dL,
  * ALT (SGPT) ≤ 2.0 × ULN (≤ 3.0 × ULN in case of liver metastases)
  * AST (SGOT) ≤ 2.0 × ULN (≤ 3.0 × ULN in case of liver metastases)
  * bilirubin ≤ 1.5 × ULN (with the exception of Gilbert's syndrome)
  * creatinine ≤ 2.0 mg/dl or 177µmol/L INR ≤ 1,5
* Patients must have the following laboratory values within normal limits or corrected to within normal limits with supplemets before the first dose of study medication:

  * Sodium
  * Potassium
  * Total calcium
* In case of patients of child bearing potential:

Negative serum pregnancy test at baseline (within 7 days prior to randomization) and agreement to remain abstinent (if it is in line with the preferred and usual lifestyle) or use single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study treatment

Exclusion criteria:

Patients will be excluded from the study for any of the following reasons:

* History of hypersensitivity reactions attributed to trastuzumab, pertuzumab, ribociclib or to other components of drug formulation
* Mandatory need for cytostatic treatment at time of study entry based on clinical judgment and national/international treatment guidelines
* Known CNS metastases
* Any concurrent severe, uncontrolled systemic disease, social or psychiatric condition that might interfere with the planned treatment and with the patient's adherence to the protocol
* Progression on prior Pertuzumab therapy
* Treatment with Pertuzumab within the last 12 months
* Prior treatment with any mTOR- or CDK4/6-inhibitor
* Treatment with any other investigational agents during trial
* Known hypersensitivity to lecithin (soya) or peanuts
* Life expectancy < 6 months
* Patients with pre-existing grade ≥2 peripheral neuropathy are excluded from taxane-based chemotherapy
* History of serious cardiac disease, including but not confined to:

  * history of documented heart failure or systolic dysfunction (LVEF < 50%)
  * high-risk uncontrolled arrhythmias i.e., atrial tachycardia with a heart rate ≥100/min at rest, significant ventricular arrhythmia (ventricular tachycardia) or higher-grade AV-block (second degree AV-block Type 2 [Mobitz 2] or third degree AV-block)
  * angina pectoris requiring anti-anginal medication
  * clinically significant valvular heart disease
  * evidence of transmural infarction on ECG
  * poorly controlled hypertension (e.g., systolic >180 mm Hg or diastolic >100 mm Hg)
  * any other cardiac condition, which in the opinion of the treating physician would make this protocol unreasonably hazardous for the patient
* Dyspnea at rest or other diseases that require continuous oxygen therapy
* Patients with poorly controlled diabetes or with evidence of clinically significant diabetic vascular complications
* Patients with known infection with HIV, hepatitis B virus, or hepatitis C virus
* Male patients
* Pregnant, lactating or women of childbearing potential without a negative pregnancy test (serum) within 7 days prior to randomization, irrespective of the method of contraception used
* Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
* Participation in another clinical study within the 30 days before registration
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 3 - 9 weeks
  safety of a dual HER2-targeted therapy with Herceptin® (trastuzumab), Perjeta® (pertuzumab) and Kisqali® (riobciclib) plus endocrine therapy as compared to a dual HER2-targeted therapy with Herceptin® (trastuzumab) and Perjeta® (pertuzumab) plus chemotherapy (followed by endocrine therapy plus ribociclib in combination with trastuzumab and pertuzumab as maintenance therapy) by the proportion of patients experiencing any adverse event (as defined by the modified adverse event score)

SECONDARY OUTCOMES:
quality-adjusted survival | 3 - 9 weeks
  to assess quality-adjusted survival (as assessed by the Q-TWiST method) and to compare it between the two treatment arms
overall response rate (ORR) | 3 - 9 weeks
  compare efficacy between the two treatment arms as assessed by overall response rate (ORR)
incidence of central nervous system (CNS) metastases and their control rate | 3 - 9 weeks
  assess the incidence of CNS metastases and control rate of preexisting CNS metastases
Analysis of Quality of life | 3 - 9 weeks
  assess additional aspects of quality of life based on the evaluation of the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) QLQ-C30 and QLQ-BR23 questionnaires
presence and number of circulating tumor cell (CTC) at different time points | 6 weeks
  determine presence and number of CTC in the peripheral blood at baseline and at different time points after the start of palliative treatment including the time of progression, and to assess the value of CTCs as indicator for therapy success
Evaluation of all reported events and all grades in both treatment arms (chemotherapy and endocrine therapy) | 3 - 9 weeks
  All reported events with all grades for evaluation of safety and tolerability of the study treatments and to to evaluate and compare toxicity of chemotherapy arm vs. endocrine treatment arm
disease control rate (DCR) | 3 - 9 weeks
  compare efficacy between the two treatment arms as assessed by disease control rate (DCR)
progression-free survival (PFS) | 3 - 9 weeks
  compare efficacy between the two treatment arms as assessed by progression-free survival (PFS)
overall survival (OS) | 3 - 9 weeks
  compare efficacy between the two treatment arms as assessed by overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Huober, MD PhD, Principal Investigator — Studienzentrale Dpt. Gyn/OB University Ulm
Locations (1):
- University Hospital Ulm Gynecology/Obstetrics, Ulm, Germany

REFERENCES:
- See also: The DETECT study concept — http://www.detect-studien.de